CLINICAL TRIAL: NCT03044236
Title: Effect of a Novel Stretching Technique on Shoulder Range of Motion and Maximum Voluntary Contraction in Overhead Athletes With Glenohumeral Internal Rotation Deficits: A Randomized Control Trial
Brief Title: Effect of a Novel Stretching Technique on Shoulder Range of Motion and Voluntary Contraction in Overhead Athletes With Glenohumeral Internal Rotation Deficits "GIRD"
Acronym: GIRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Everett Lohman, Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5170032
Record Dates: First submitted 2017-01-30; First posted 2017-02-06 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2018-08

CONDITIONS: Glenohumeral Internal Rotation Deficits

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel Stretching Technique (Experimental): Participants will perform the novel stretch in a supine position. Participants will place a small ball between their knees and squeeze the ball. Participants will be then bridge as high as possible . Participants will then flex their shoulder and elbow to 90°, and actively rotate to the end of ROM. Participants will use the other hand to push to the point of mild discomfort and simultaneously maintain contraction while progressing the stretch.
  Interventions: Procedure: Stretching
- Traditional Stretching Technique (Active Comparator): Participants will perform the modified sleeper stretch in a side-lying position on the side of the throwing shoulder with the throwing shoulder and elbow flexed to 90° . The participants will be instructed to allow the throwing shoulder to naturally fall into internal rotation to the end ROM where resistance will be felt . The participants will be then instructed to use the non-throwing hand to push the throwing shoulder into further internal rotation to the point of mild discomfort by applying pressure at the area of the wrist joint.
  Interventions: Procedure: Stretching

INTERVENTIONS:
Procedure: Stretching — The novel stretching technique will be done on a supine position. subjects will be asked bridge as high as possible. After That, Participants will then flex their shoulder and elbow to 90°. Participants will use the other hand to push to the point of mild discomfort and simultaneously maintain contraction while progressing the stretch.

SUMMARY:
To examine and compare the effect of a novel stretching technique and traditional stretching on glenohumeral range of motion, strength, maximum voluntary contraction, pain, and subject satisfaction in overhead athletes with glenohumeral internal rotation deficits through a randomized clinical study.

DETAILED DESCRIPTION:
To examine and compare the effect of a novel stretching technique and traditional stretching on glenohumeral range of motion, strength, maximum voluntary contraction, pain, and subject satisfaction in overhead athletes with glenohumeral internal rotation deficits through a randomized clinical study. The investigators hypothesize that this type of novel intervention will help subjects with GIRD to restore range of motion, experience less pain and maintain the strength and motor unit recruitment following the novel intervention. This will help us to assess the potential beneficial effect of such intervention and to fill the gap in knowledge and help health care professionals to adequately select the right treatment modality.

Independent Variable

1. Type of Intervention:

* Traditional Stretching (Modified Sleep Stretch). VS
* Novel Stretching (Active Shoulder Internal Rotation while Bridging) 2. Time
* Pre VS post intervention Dependent Variables

  1. Glenohumeral internal rotation ROM
  2. Maximal glenohumeral external rotation isometric strength.
  3. Mean motor unit recruitment (EMG) of the glenohumeral external rotator (infraspinatus) and internal rotators (pectoralis major and latissumus dorsi)
  4. Pain
  5. Subject satisfaction

Instrumentation :

1. Glenohumeral internal & external rotation ROM: will be measured at baseline and at week four-post intervention for all participants. We will use the digital inclinometer. Research by (Kolber et al.,2011 ) showed this instrument to be reliable with an intra-rater ICC =0.87 and inter-rater ICC =0.93
2. Electronic push/pull dynamometer: At the end feel ROM, and before ROM is measured, the therapist will apply the same amount of pressure to all subjects to ensure reliable/ valid ROM measurements.
3. Maximal Glenohumeral External Rotation Isometric Strength will be measured using a MicroFET2 handheld digital dynamometer. This device was shown to be reliable with an intra-rater ICC =0.85 and inter-rater ICC =0.85.
4. Maximum Voluntary Contraction: will be measured using a 44 Delsys Bagnoli portable surface electromyography (sEMG) system.
5. Pain: will be measured using the Numeric Pain Rating Scale (NPRS). The NPRS has shown to have a valid, reliable and appropriate for use in clinical practice

Procedures:

All participants will perform the static stretching (SS) conditions by themselves. The two stretching techniques will be home-based program.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the age of 18 and 45.
* Perform overhead sports activities in the past 3 months.
* Participants are required to display ≥ 20° less glenohumeral internal rotation ROM in their dominant shoulder compare to the non- dominate shoulder.
* Participants will be included with or without pain during shoulder activities.

Exclusion Criteria:

* Will exclude participants who are still recovering from previous surgery of the shoulder and elbow complex in the past 3 months, and currently receiving medical intervention for the shoulder.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Glenohumeral internal rotation ROM | Change from baseline at week 4
  The investigators will use the digital inclinometer

SECONDARY OUTCOMES:
Maximal glenohumeral external rotation isometric strength | Change from baseline at week 4
  will be measured using a MicroFET2 handheld digital dynamometer

OTHER OUTCOMES:
Mean motor unit recruitment (EMG) of the glenohumeral external rotator (infraspinatus) and internal rotators (pectoralis major and latissumus dorsi) | Change from baseline at week 4
  will be measured using surface electromyography (sEMG) system
Pain will be measured using the Numeric Pain Rating Scale | Change from baseline at week 4
  will be measured using the Numeric Pain Rating Scale
Subject satisfaction will be measured using the Subject satisfaction Form | Week 4
  will be measured using the Subject satisfaction Form

CONTACTS AND LOCATIONS:
Overall Officials: Everett Lohman, DSc, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda U, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gharisia O, Lohman E, Daher N, Eldridge A, Shallan A, Jaber H. Effect of a novel stretching technique on shoulder range of motion in overhead athletes with glenohumeral internal rotation deficits: a randomized controlled trial. BMC Musculoskelet Disord. 2021 Apr 30;22(1):402. doi: 10.1186/s12891-021-04292-8. PMID 33941143